CLINICAL TRIAL: NCT04733820
Title: Clinical Efficacy of Adjuvant Chemotherapy in Patients With Locally Advanced Cervical Cancer Who Did Not Meet the NCCN Guidelines for Adjuvant Treatment After NACT Combined With Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Women's Hospital School Of Medicine Zhejiang University (Other); Qilu Hospital of Shandong University (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Hunan Cancer Hospital (Other); The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Ding Ma, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-S111
Record Dates: First submitted 2021-01-21; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Uterine Cervical Neoplasms; Cervical Cancer
Keywords: Cervical Cancer; NACT; Adjuvant Chemotherapy; Locally Advanced Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant chemotherapy group (Experimental): Participant will receive at least 2 cycles of adjuvant chemotherapy. If having any of the following factors, participant will receive additional 2 cycles of adjuvant chemotherapy per risk factor. All patients received maximum 6 cycles of postoperative chemotherapy.
  Risk factors: (1) Deep cervical invasion（≥ 2/3）；（2）Differentiation grade 2-3；（3）Lymphatic vascular space infiltration；（4）Adenocarcinoma or adenosquamous carcinoma；（5）Tumor size ≥ 4cm before surgery.
  Interventions: Drug: Adjuvant chemotherapy
- Control group (No Intervention): The participants receive no intervention.

INTERVENTIONS:
Drug: Adjuvant chemotherapy — Drug: Paclitaxel or docetaxel + Cisplatin or carboplatin Paclitaxel 135-175mg/m2 over 3 hours or docetaxel 70-75 mg/m2， 30min ＋ Cisplatin 75-80mg/m2 or carboplatin AUC = 5, repeat per 21 days.
  Arms: Adjuvant chemotherapy group

SUMMARY:
This is a prospective, phase 3 randomized controlled clinical trial. Cervical cancer patients with FIGO stage IB3, Ⅱ A2 or IIB with tumor size> 4 cm will be enrolled. Patients will undergo 2-3 cycles of neoadjuvant chemotherapyradical (NACT) followed by laparotomic or laparoscopic hysterectomy + pelvic lymphadenectomy with cervical cancer foci sealed before dissection of the vagina and without uterine manipulator. Patients meet criteria of adjuvant therapy according to NCCN guideline after surgery will be weeded out, and who do not meet criteria of adjuvant therapy will be randomly selected to undergo adjuvant chemotherapy or just follow-up visit. The primary endpoint was disease-free survival (DFS) rate at 5 year. The secondary endpoints were 5-year overall survival (OS), safety and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical stage IB3-IIB cervical cancer (FIGO, 2018 standard) with the tumor diameter > 4cm before treatment.
2. Pathologically confirmed cervical cancer, including cervical squamous cell carcinoma, adenocarcinoma and adenosquamous carcinoma.
3. Age：18-70 years old.
4. ECOG status score ≤1;
5. WBC≥3.5*10^9/L, NEU≥1.5*10^9/L, Platelet≥80×10^9 /L; AST and ALT ≤1.5 times normal upper limit; Total bilirubin ≤1.5 times the upper limit of normal value; serum creatinine and blood urea nitrogen ≤the upper limit of normal value.
6. Well-compliance and willing to keep in touch.
7. Able to sign informed consent, including complying with the requirements and restrictions listed in the Informed Consent (ICF) and this protocol.

Exclusion Criteria:

1. After 2-3 cycles of neoadjuvant chemotherapy, patients do not undergo laparotomic or laparoscopic extensive hysterectomy + pelvic lymph node dissection with cervical cancer foci sealed before dissection of the vagina and without uterine manipulator.
2. Neoadjuvant chemotherapy regimens are different from postoperative adjuvant therapy regimens.
3. Postoperative high risk factors: ① lymph node metastasis, ② parauterine infiltration, ③ positive surgical margin.
4. Postoperative risk factors meet the Sedlis standard of the NCCN guideline.
5. Participate in other clinical trials.
6. Severe diseases of other important systems and organs.
7. Persons without disposing capacity.
8. Drug and/or alcohol abuse.
9. Unable or unwilling to sign informed consents.
10. Not eligible for the study judged by researchers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 5 year
  DFS is defined as the time interval between the date of random assignment and the date of the first documented evidence of relapse at any site or death related to cancer (including toxicity), whichever occurred first.

SECONDARY OUTCOMES:
Overall survival （OS） | 5 year
  OS is defined as the time from the date of randomization until death of any cause.
Quality of Life Outcomes | 5 years
  Patients are asked to complete the questionnaire EORTC QLQ-C30
Quality of Life Outcomes of cervical cancer | 5 years
  Patients are asked to complete the questionnaire EORTC QLQ-CX24
Incidence of Toxicity | 5 years
  The toxicity induced by chemotherapy during observation time will be estimated on the basis of the National Cancer Institute Common Toxicity Criteria Version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided